CLINICAL TRIAL: NCT03901586
Title: Satisfaction and Long-term Anatomic Efficacy Study on Patients Who Underwent a Richter Intervention in the Obstetric and Gynecology Department of Foch Hospital Since 2008
Acronym: RICHTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018_0072
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2018-11

CONDITIONS: Genital Prolapse
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients who had Richter intervention (Experimental)
  Interventions: Other: Satisfaction assessment; Other: Quality of life; Other: Gynecological assessment

INTERVENTIONS:
Other: Satisfaction assessment — Patient will be asked to assess their satisfaction concerning the Richter procedure and its long term effect
Other: Quality of life — The Quality of life will be assessed with 3 questionnaires (I-Qol / PISQ-12/PFDI-20)
Other: Gynecological assessment — An optional gynecological consult is proposed to the patients to better estimate the gynecological long-term impact of the procedure

SUMMARY:
Satisfaction and Long-term Anatomic Efficacy will be assessed on Patients Who Underwent a Richter Intervention in the Obstetric and Gynecology Department of Foch Hospital Since 2008.

DETAILED DESCRIPTION:
Satisfaction and Long-term Anatomic Efficacy will be assessed on Patients Who Underwent a Richter Intervention in the Obstetric and Gynecology Department of Foch Hospital Since 2008.

ELIGIBILITY:
Inclusion Criteria:

* Patient who underwent a Richter intervention between 01/01/2008 and 31/12/2017 in the Gynecology Department of Foch Hospital

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Long-term satisfaction of the Richter procedure | 4 months
  It will be ask to the patients to evaluate their satisfaction of the procedure, base on a 4-answer scale ("Not at all satisfied", "Not very satisfied", "Moderately satisfied", "Fully satisfied")

SECONDARY OUTCOMES:
Long term anatomic impact of the procedure | 7 months
  An optional gynecological consult is proposed to the patients
Post-operative complications | 7 months
  Post-operative complications will be collected and compared to the anatomic impact of the procedure and the patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Angeline Favre-Inhofer, Principal Investigator — Hôpital Foch; Jean-Marc Ayoubi, Study Director — Hôpital Foch
Locations (1):
- Hôpital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No